CLINICAL TRIAL: NCT04015518
Title: Multi-center, Double-blind, Randomised, Placebo-controlled, Phase IIb Dose-finding Study to Evaluate Safety and Efficacy of Different Subcutaneous Doses of BI 655130 in Patients With Moderate to Severe Palmoplantar Pustulosis (PPP)
Brief Title: A Study to Test How Effective and Safe Different Doses of BI 655130 Are in Patients With a Moderate to Severe Form of the Skin Disease Palmoplantar Pustulosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1368-0016; 2018-003078-28 (EudraCT Number)
Record Dates: First submitted 2019-07-09; First posted 2019-07-11 (Actual); Results first posted 2022-07-28 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Palmoplantar Pustulosis (PPP)
MeSH Terms: conditions — Psoriasis | interventions — spesolimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Placebo & Spesolimab (Other): Subcutaneous injections of placebo matching Spesolimab, with subcutaneous injections of Spesolimab starting at week 16, for a total treatment time of 52 weeks.
  Interventions: Drug: Spesolimab; Drug: Placebo
- Spesolimab 'Speso Low' (Experimental): Subcutaneous injections of Spesolimab in a low dose scheme for a total treatment time of 52 weeks.
  Interventions: Drug: Spesolimab
- Spesolimab 'Speso Medium-low' (Experimental): Subcutaneous injections of Spesolimab in a medium-low dose scheme for a total treatment time of 52 weeks.
  Interventions: Drug: Spesolimab
- Spesolimab 'Speso Medium-high' (Experimental): Subcutaneous injections of Spesolimab in a medium-high dose scheme for a total treatment time of 52 weeks.
  Interventions: Drug: Spesolimab
- Spesolimab 'Speso High' (Experimental): Subcutaneous injections of Spesolimab in a high dose scheme for a total treatment time of 52 weeks.
  Interventions: Drug: Spesolimab

INTERVENTIONS:
Drug: Spesolimab — Subcutaneous injections of Spesolimab starting at week 16, for a total treatment time until week 52.
  Arms: Placebo & Spesolimab
Drug: Placebo — Subcutaneous injections of placebo matching Spesolimab from week 0 to 16.
  Arms: Placebo & Spesolimab
Drug: Spesolimab — Subcutaneous injections of Spesolimab in a low dose scheme for a total treatment time of 52 weeks.
  Arms: Spesolimab 'Speso Low'
Drug: Spesolimab — Subcutaneous injections of Spesolimab in a medium-low dose scheme for a total treatment time of 52 weeks.
  Arms: Spesolimab 'Speso Medium-low'
Drug: Spesolimab — Subcutaneous injections of Spesolimab in a medium-high dose scheme for a total treatment time of 52 weeks.
  Arms: Spesolimab 'Speso Medium-high'
Drug: Spesolimab — Subcutaneous injections of Spesolimab in a high dose scheme for a total treatment time of 52 weeks.
  Arms: Spesolimab 'Speso High'

SUMMARY:
The primary objective is to provide dose-ranging data for 4 dose regimens of BI 655130 compared to placebo on the primary endpoint of percentage change from baseline in PPP ASI at Week 16. The target dose(s) will be estimated from the model by incorporating information on the minimum clinically relevant effect and accounting for safety.

Supportive dose-ranging assessments will also be done on pre-specified secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years of legal age (according to local legislation) at screening.
* Diagnosis of Palmoplantar Pustulosis defined as presence of primary, persistent (>3 months duration), sterile, macroscopically visible pustules on the palms and/or soles, without or with plaque psoriasis elsewhere on the body.
* PPP PGA of at least moderate severity (≥3) at screening and baseline.
* A minimum PPP ASI score of 12 at screening and baseline.
* Male or female patients. Women of childbearing potential (WOCBP) must be ready and able to use highly effective methods of birth control per ICH M3 (R2).
* Signed and dated written informed consent in accordance with ICH GCP and local legislation prior to admission to the trial.
* Further criteria apply.

Exclusion Criteria:

* Women who are pregnant, nursing, or who plan to become pregnant while in the trial.
* Severe, progressive, or uncontrolled condition such as renal, hepatic, haematological, endocrine, pulmonary, cardiac, neurologic, cerebral, or psychiatric disease, or signs and symptoms thereof.
* Presence or known history of anti-TNF-induced PPP-like disease.
* Patient with a transplanted organ (with exception of a corneal transplant >12 weeks Prior to screening) or who have ever received stem cell therapy (e.g., Prochymal).
* Known history of lymphoproliferative disease, including lymphoma, or signs and symptoms suggestive of possible lymphoproliferative disease, such as lymphadenopathy and/or splenomegaly.
* Further criteria apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2020-08-06 (Actual); Study Completion 2021-07-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (88):
- United States (14):
  - Total Skin and Beauty Dermatology Center, PC, Birmingham, Alabama
  - Wallace Medical Group, Beverly Hills, California
  - Therapeutics Clinical Research, San Diego, California
  - Advanced Medical Research PC, Sandy Springs, Georgia
  - Epiphany Dermatology of Kansas, LLC, Overland Park, Kansas
  - University of Missouri Health System, Columbia, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Skin Specialists, P.C., Omaha, Nebraska
  - The Psoriasis Treatment Center of Central New Jersey, East Windsor, New Jersey
  - Paddington Testing Co., Inc., Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Menter Dermatology Research Institute, Dallas, Texas
  - University of Utah Health, Murray, Utah
  - Virginia Clinical Research, Inc., Norfolk, Virginia
- Australia (5):
  - Paratus Clinical Research Woden, Phillip, Australian Capital Territory
  - Westmead Hospital, Westmead, New South Wales
  - Veracity Clinical Research, Wooloongabba, Queensland
  - Skin Health Institute Inc, Carlton, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Belgium (2):
  - Brussels - UNIV Saint-Luc, Brussels
  - UZ Leuven, Leuven
- Canada (7):
  - CARe Clinic, Red Deer, Alberta
  - Dr. Irina Turchin PC Inc., Fredericton, New Brunswick
  - SimcoDerm Medical and Surgical Dermatology Centre, Barrie, Ontario
  - The Guenther Dermatology Research Centre, London, Ontario
  - York Dermatology Clinic and Research Centre, Richmond Hill, Ontario
  - K. Papp Clinical Research Inc., Waterloo, Ontario
  - Innovaderm Research Inc., Montreal, Quebec
- Czechia (3):
  - CCBR Czech a.s., Pardubice
  - Sanatorium Prof. Arenebergera, Prague
  - CCBR Czech Prague s.r.o., Prague
- France (3):
  - HOP l'Archet, Nice
  - HOP Saint-Louis, Paris
  - HOP Larrey, Toulouse
- Germany (5):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsklinikum Frankfurt, Frankfurt am Main
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel
- Hungary (4):
  - CRU Hungary Ltd, Private Practice, Miskolc, Miskolc
  - University of Pecs, Pécs
  - Markusovszky University Teaching Hospital, Szombathely
  - Veszprem County Csolnoky Ferenc Hospital, Veszprém
- Japan (30):
  - Nagoya City University Hospital, Aichi, Nagoya
  - Fujita Health University Hospital, Aichi, Toyoake
  - Tokyo Dental College Ichikawa General Hospital, Chiba, Ichikawa
  - Ehime University Hospital, Ehime, Toon
  - Fukuoka University Hospital, Fukuoka, Fukuoka
  - Gifu University Hospital, Gifu, Gifu
  - Asahikawa Kosei General Hospital, Hokkaido, Asahikawa
  - Asahikawa Medical University Hospital, Hokkaido, Asahikawa
  - Takagi Dermatological Clinic, Hokkaido, Obihiro
  - Hosui General Medical Clinic, Hokkaido, Sapporo
  - Takamatsu Red Cross Hospital, Kagawa, Takamatsu
  - Sagamihara National Hospital, Kanagawa, Sagamihara
  - Kumamoto University Hospital, Kumamoto, Kumamoto
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto, Kyoto
  - Tohoku University Hospital, Miyagi, Sendai
  - Shinshu University Hospital, Nagano, Matsumoto
  - Okayama University Hospital, Okayama, Okayama
  - University of the Ryukyus Hospital, Okinawa, Nakagami-gun
  - Kindai University Hospital, Osaka, Osaka-sayama
  - Nakatsu Dermatology Clinic, Osaka, Osaka
  - Osaka City University Hospital, Osaka, Osaka
  - Osaka University Hospital, Osaka, Suita
  - Shiga University of Medical Science Hospital, Shiga, Otsu
  - Jichi Medical University Hospital, Tochigi, Shimotsuke
  - Teikyo University Hospital, Tokyo, Itabashi-ku
  - Nihon University Itabashi Hospital, Tokyo, Itabashi-ku
  - Tokyo Medical University Hospital, Tokyo, Shinjuku-ku
  - Seibo Hospital, Tokyo, Shinjuku
  - Shirasaki Dermatology and Neurology Clinic, Toyama, Takaoka
  - Wakayama Medical University Hospital, Wakayama, Wakayama
- Amphia Ziekenhuis, Breda, Netherlands
- Poland (5):
  - Barbara Rewerska Diamond Clinic, Krakow, Krakow
  - Dermoklinika medical center, Lodz, Lodz
  - Independent Public Clin.Hosp.no1 Lublin, Lublin
  - Municipal Hospital Complex in Olsztyn, Olsztyn
  - Dermmedica Sp. z o.o., Wroclaw, Wroclaw
- Russia (3):
  - SBHI Chelyabinsk Reg.Clin.Derma.Dispen., Chelyabinsk
  - LLC "Medical Center Azbuka Zdorovia", Kazan'
  - Dermatovenereological Dispensary #10, St. Petersburg, Saint Petersburg
- South Korea (3):
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul
- National Taiwan University Hospital, Taipei, Taiwan
- United Kingdom (2):
  - Royal Devon and Exeter Hospital, Exeter
  - Guy's Hospital, London

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- [Derived] Lebwohl MG, Thoma C, Haeufel T. Spesolimab use in generalised pustular psoriasis flares - Authors' reply. Lancet. 2024 Aug 31;404(10455):847-848. doi: 10.1016/S0140-6736(24)01557-5. No abstract available. PMID 39216969
- [Derived] Burden AD, Bissonnette R, Navarini AA, Murakami M, Morita A, Haeufel T, Ye B, Baehner F, Terui T. Spesolimab Efficacy and Safety in Patients with Moderate-to-Severe Palmoplantar Pustulosis: A Multicentre, Double-Blind, Randomised, Placebo-Controlled, Phase IIb, Dose-Finding Study. Dermatol Ther (Heidelb). 2023 Oct;13(10):2279-2297. doi: 10.1007/s13555-023-01002-1. Epub 2023 Sep 20. PMID 37731086
- See also: Related Info — http://mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomised, placebo-controlled, double-blind, parallel-design trial comparing 5 treatment arms over 52 weeks. Randomisation was stratified for Japan versus non-Japan. Patients who completed the treatment period without premature discontinuation and obtained an individual health benefit, per investigator judgement, could continue treatment with spesolimab in the open-label extension trial 1368-0024.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Overall Study
Arm/Group | Placebo & Spesolimab | Spesolimab 'Speso Low' | Spesolimab 'Speso Medium-low' | Spesolimab 'Speso Medium-high' | Spesolimab 'Speso High'
Started | 43 | 22 | 21 | 22 | 44
Full Analysis Set (FAS) | 43 | 22 | 21 | 22 | 44
Completed | 32 | 19 | 18 | 17 | 32
Not Completed | 11 | 3 | 3 | 5 | 12
Not completed — Adverse Event | 6 | 1 | 1 | 3 | 3
Not completed — Lack of Efficacy | 1 | 0 | 1 | 0 | 4
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1 | 1
Not completed — Patient did not come for consecutive visits | 0 | 1 | 0 | 0 | 0
Not completed — not willing to travel due to Covid-19 | 0 | 0 | 1 | 0 | 0
Not completed — Patient wants to discontinue treatment | 0 | 0 | 0 | 1 | 0
Not completed — Difficult for patient to come to the hospital | 0 | 0 | 0 | 0 | 1
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 1
Not completed — Personal reasons | 1 | 0 | 0 | 0 | 1
Not completed — Withdrew consent | 1 | 0 | 0 | 0 | 0
Not completed — Prostate carcinoma | 1 | 0 | 0 | 0 | 0
Not completed — Could not keep appointments due to work | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAF): This patient set includes all patients who were randomised and received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo & Spesolimab | Spesolimab 'Speso Low' | Spesolimab 'Speso Medium-low' | Spesolimab 'Speso Medium-high' | Spesolimab 'Speso High' | Total
Number analyzed (Participants) | 43 | 22 | 21 | 22 | 44 | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (10.1) | 54.2 (12.3) | 51.6 (7.9) | 52.8 (9.2) | 53.4 (13.0) | 54.4 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 15 | 16 | 17 | 27 | 110
  Male | 8 | 7 | 5 | 5 | 17 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 40 | 20 | 19 | 21 | 41 | 141
  Unknown or Not Reported | 3 | 2 | 2 | 1 | 3 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 18 | 9 | 9 | 9 | 15 | 60
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 0 | 1
  White | 21 | 11 | 10 | 12 | 26 | 80
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 2 | 1 | 3 | 11
Palmoplantar Pustulosis Area and Severity Index (PPP ASI) [Mean (Standard Deviation); unit: Score on a scale] — The PPP ASI is an investigator assessment of the extent and severity of pustular and plaque lesions on the palms and soles presenting in PPP patients. This tool provides a numeric scoring for patients overall PPP disease state, ranging from 0 (best) to 72 (worst). It is a linear combination of the percent of surface area of skin that is affected on the palms and soles of the body and the severity of erythema, pustules, and scaling (desquamation).
  Score on a scale | 27.07 (12.44) | 23.85 (9.42) | 23.62 (11.02) | 26.65 (11.20) | 24.00 (10.25) | 25.18 (11.00)

OUTCOME MEASURES:

1. Primary Outcome: The Percentage Change in Palmoplantar Pustulosis Area and Severity Index (PPP ASI) at Week 16 From Baseline
Description: The percentage change in PPP ASI at Week 16 from baseline. The PPP ASI is a tool that provides a numeric scoring for patients overall PPP disease state, ranging from 0 (best) to 72 (worst). It is a linear combination of the percent of surface area of skin that is affected on the palms and soles of the body and the severity of erythema, pustules, and scaling (desquamation): The percent change from baseline is calculated as (PPP ASI current - PPP ASI baseline) / PPP ASI baseline * 100%.
  Least square (LS) means, differences and confidence intervals were estimated by (Restricted maximum likelihood)-based Mixed effect model for repeated measurements (MMRM) including the fixed, categorical effects of treatment at each visit, region and the continuous effect of baseline at each visit as well as random effects of subject. Values post rescue medication or 6 weeks following last study treatment before discontinuation were censored. Unstructured covariance matrix was used.
Time Frame: week 0 (baseline) and week 16
Population: Full Analysis Set (FAS): This patient set includes all patients who were randomised and received at least one dose of study drug. Only subjects with non missing endpoint data were included.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of change in PPP ASI
Arm/Group | Placebo | Spesolimab 'Speso Low' | Spesolimab 'Speso Medium-low' | Spesolimab 'Speso Medium-high' | Spesolimab 'Speso High'
Number analyzed (Participants) | 38 | 20 | 21 | 20 | 41
Percentage of change in PPP ASI | -33.6 [-43.5 to -23.7] | -44.2 [-57.8 to -30.6] | -48.3 [-61.8 to -34.7] | -46.2 [-59.9 to -32.6] | -38.9 [-48.5 to -29.3]
Statistical Analysis 1: Comparison: Placebo vs Spesolimab 'Speso Low'; Test type: Other — Mixed-effects Model Repeated Measures (MMRM) estimates were used as input for the MCP-Mod. MMRM included'baseline' as a continuous covariate, and 'visit', 'treatment', 'region' (stratification according to Japan vs. non-Japan), 'visit*treatment' and 'visit*baseline' interaction as fixed effects as well as the random 'subject' effect. Covariance structure= Unstructured; p = 0.2179, Mixed Models Analysis; Kenward-Roger was used to estimate denominator degrees of freedom; Difference of adjusted means = -10.5, 95% CI 2-sided [-27.4 to 6.3], Standard Error of Mean 8.5 — Difference was calculated as Speso - placebo
Statistical Analysis 2: Comparison: Placebo vs Spesolimab 'Speso Medium-low'; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0883, Mixed Models Analysis; Kenward-Roger was used to estimate denominator degrees of freedom; Difference of adjusted means = -14.6, 95% CI 2-sided [-31.5 to 2.2], Standard Error of Mean 8.5 — Difference was calculated as Speso - placebo
Statistical Analysis 3: Comparison: Placebo vs Spesolimab 'Speso Medium-high'; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.1414, Mixed Models Analysis; Kenward-Roger was used to estimate denominator degrees of freedom; Difference of adjusted means = -12.6, 95% CI 2-sided [-29.4 to 4.3], Standard Error of Mean 8.5 — Difference was calculated as Speso - placebo
Statistical Analysis 4: Comparison: Placebo vs Spesolimab 'Speso High'; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.4514, Mixed Models Analysis; Kenward-Roger was used to estimate denominator degrees of freedom; Difference of adjusted means = -5.3, 95% CI 2-sided [-19.1 to 8.6], Standard Error of Mean 7.0 — Difference was calculated as Speso - placebo
Statistical Analysis 5: Comparison: Placebo vs Spesolimab 'Speso Low' vs Spesolimab 'Speso Medium-low' vs Spesolimab 'Speso Medium-high' vs Spesolimab 'Speso High'; A flat vs. non-flat dose-response relationship across the 4 doses of Spesolimab and placebo was tested using the Multiple Comparison Procedure - Modelling (MCP-Mod) approach which evaluated simultaneously 5 different plausible dose-response patterns (linear, Emax, exponential, logistic, Sigmoid Emax) while protecting the overall probability of type I error (one-sided alpha of 0.05); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.2120, MCP-Mod linear model fit — Adjusted for multiplicity
Statistical Analysis 6: Comparison: Placebo vs Spesolimab 'Speso Low' vs Spesolimab 'Speso Medium-low' vs Spesolimab 'Speso Medium-high' vs Spesolimab 'Speso High'; [analysis description as in outcome 1, analysis 5]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.1057, MCP-Mod Emax model fit — Adjusted for multiplicity; Assumed 70% of the maximum effect was achieved at the "low dose" regimen
Statistical Analysis 7: Comparison: Placebo vs Spesolimab 'Speso Low' vs Spesolimab 'Speso Medium-low' vs Spesolimab 'Speso Medium-high' vs Spesolimab 'Speso High'; [analysis description as in outcome 1, analysis 5]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.5241, MCP-Mod Exponential model fit — Adjusted for multiplicity; Assumed 25% of the maximum effect was achieved at the "medium-low dose" regimen
Statistical Analysis 8: Comparison: Placebo vs Spesolimab 'Speso Low' vs Spesolimab 'Speso Medium-low' vs Spesolimab 'Speso Medium-high' vs Spesolimab 'Speso High'; [analysis description as in outcome 1, analysis 5]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.2773, MCP-Mod Logistic model fit — Adjusted for multiplicity; Assumed 20% of maximum effect was achieved at the "low dose", 95% of maximum effect was achieved at "medium high dose"
Statistical Analysis 9: Comparison: Placebo vs Spesolimab 'Speso Low' vs Spesolimab 'Speso Medium-low' vs Spesolimab 'Speso Medium-high' vs Spesolimab 'Speso High'; [analysis description as in outcome 1, analysis 5]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.3867, MCP-Mod Sigmoid Emax model fit — Adjusted for multiplicity; Assumed 10% of the maximum effect was achieved at "low dose", 80% of the maximum effect was achieved at the "medium-high dose"

2. Secondary Outcome: Change From Baseline in Palmoplantar Pustulosis Pain Visual Analogue Scale (VAS) Score at Week 4
Description: Change from baseline in Palmoplantar Pustulosis Pain Visual Analogue Scale (VAS) score at Week 4. The PPP Pain VAS is a unidimensional measure of pain intensity due to palmoplantar pustulosis on palms and/or soles. It is a continuous scale comprised of a horizontal or vertical line, 10 centimeters (cm) in length, anchored by word descriptors at each end (score ranges from "no pain" at 0 cm to "very severe pain" at 10 cm). The patient was asked to place a vertical ( | ) mark on the horizontal line to indicate the severity of the pain.
  Least square (LS) means, differences and confidence intervals were estimated by (Restricted maximum likelihood)-based MMRM including the fixed, categorical effects of treatment at each visit, region and the continuous effect of baseline at each visit as well as random effects of subject. Values post rescue medication or 6 weeks following last study treatment before discontinuation were censored. Unstructured covariance matrix was used.
Time Frame: week 0 (baseline) and week 4.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Groups:
- Placebo: Subcutaneous injection of placebo matching Spesolimab 150 milligram (mg)/syringe, Loading period with 4 injections per visit (weekly up to Week 4).
Arm/Group | Placebo | Spesolimab 'Speso Low' | Spesolimab 'Speso Medium-low' | Spesolimab 'Speso Medium-high' | Spesolimab 'Speso High'
Number analyzed (Participants) | 38 | 20 | 21 | 20 | 41
Score on a scale | -9.3 [-17.0 to -1.6] | -15.4 [-26.1 to -4.8] | -14.7 [-25.7 to -3.8] | -12.8 [-23.5 to -2.1] | -18.7 [-26.3 to -11.1]
Statistical Analysis 1: Comparison: Placebo vs Spesolimab 'Speso Low'; Test type: Other — [test comment as in outcome 1, analysis 1]; Difference of adjusted means = -6.1, 95% CI 2-sided [-19.3 to 7.1], Standard Error of Mean 6.7 — Difference was calculated as Speso - placebo
Statistical Analysis 2: Comparison: Placebo vs Spesolimab 'Speso Medium-low'; Test type: Other — [test comment as in outcome 1, analysis 1]; Difference of adjusted means = -5.4, 95% CI 2-sided [-18.8 to 8.0], Standard Error of Mean 6.8 — Difference was calculated as Speso - placebo
Statistical Analysis 3: Comparison: Placebo vs Spesolimab 'Speso Medium-high'; Test type: Other — [test comment as in outcome 1, analysis 1]; Difference of adjusted means = -3.5, 95% CI 2-sided [-16.6 to 9.7], Standard Error of Mean 6.6 — Difference was calculated as Speso - placebo
Statistical Analysis 4: Comparison: Placebo vs Spesolimab 'Speso High'; Test type: Other — [test comment as in outcome 1, analysis 1]; Difference of adjusted means = -9.4, 95% CI 2-sided [-20.3 to 1.4], Standard Error of Mean 5.5 — Difference was calculated as Speso - placebo

3. Secondary Outcome: Change From Baseline in Palmoplantar Pustulosis Pain Visual Analogue Scale (VAS) Score at Week 16
Description: Change from baseline in Palmoplantar Pustulosis Pain Visual Analogue Scale (VAS) score at Week 16. The PPP Pain VAS is a unidimensional measure of pain intensity due to palmoplantar pustulosis on palms and/or soles. It is a continuous scale comprised of a horizontal or vertical line, 10 centimeters (cm) in length, anchored by word descriptors at each end (score ranges from "no pain" at 0 cm to "very severe pain" at 10 cm). The patient was asked to place a vertical ( | ) mark on the horizontal line to indicate the severity of the pain.
  Least square (LS) means, differences and confidence intervals were estimated by (Restricted maximum likelihood)-based MMRM including the fixed, categorical effects of treatment at each visit, region and the continuous effect of baseline at each visit as well as random effects of subject. Values post rescue medication or 6 weeks following last study treatment before discontinuation were censored. Unstructured covariance matrix was used.
Time Frame: week 0 (baseline) and week 16.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Placebo | Spesolimab 'Speso Low' | Spesolimab 'Speso Medium-low' | Spesolimab 'Speso Medium-high' | Spesolimab 'Speso High'
Number analyzed (Participants) | 38 | 20 | 21 | 20 | 41
Score on a scale | -14.7 [-22.7 to -6.7] | -18.7 [-29.8 to -7.7] | -13.8 [-24.8 to -2.8] | -18.9 [-30.0 to -7.8] | -22.4 [-30.2 to -14.6]
Statistical Analysis 1: Comparison: Placebo vs Spesolimab 'Speso Low'; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.5595, Mixed Models Analysis; Kenward-Roger was used to estimate denominator degrees of freedom; Difference of adjusted means = -4.1, 95% CI 2-sided [-17.7 to 9.6], Standard Error of Mean 6.9 — Difference was calculated as Speso - placebo
Statistical Analysis 2: Comparison: Placebo vs Spesolimab 'Speso Medium-low'; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.8968, Mixed Models Analysis; Kenward-Roger was used to estimate denominator degrees of freedom; Difference of adjusted means = 0.9, 95% CI 2-sided [-12.7 to 14.5], Standard Error of Mean 6.9 — Difference was calculated as Speso - placebo
Statistical Analysis 3: Comparison: Placebo vs Spesolimab 'Speso Medium-high'; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.5456, Mixed Models Analysis; Kenward-Roger was used to estimate denominator degrees of freedom; Difference of adjusted means = -4.2, 95% CI 2-sided [-17.9 to 9.5], Standard Error of Mean 6.9 — Difference was calculated as Speso - placebo
Statistical Analysis 4: Comparison: Placebo vs Spesolimab 'Speso High'; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.1762, Mixed Models Analysis; Kenward-Roger was used to estimate denominator degrees of freedom; Difference of adjusted means = -7.7, 95% CI 2-sided [-19.0 to 3.5], Standard Error of Mean 5.7 — Difference was calculated as Speso - placebo
Statistical Analysis 5: Comparison: Placebo vs Spesolimab 'Speso Low' vs Spesolimab 'Speso Medium-low' vs Spesolimab 'Speso Medium-high' vs Spesolimab 'Speso High'; [analysis description as in outcome 1, analysis 5]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.1726, MCP-Mod linear model fit — Adjusted for multiplicity
Statistical Analysis 6: Comparison: Placebo vs Spesolimab 'Speso Low' vs Spesolimab 'Speso Medium-low' vs Spesolimab 'Speso Medium-high' vs Spesolimab 'Speso High'; [analysis description as in outcome 1, analysis 5]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.2353, MCP-Mod Emax model fit — Adjusted for multiplicity; Assumed 70% of the maximum effect was achieved at the "low dose" regimen
Statistical Analysis 7: Comparison: Placebo vs Spesolimab 'Speso Low' vs Spesolimab 'Speso Medium-low' vs Spesolimab 'Speso Medium-high' vs Spesolimab 'Speso High'; [analysis description as in outcome 1, analysis 5]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.1346, MCP-Mod Exponential model fit — Adjusted for multiplicity; Assumed 25% of the maximum effect was achieved at the "medium-low dose" regimen
Statistical Analysis 8: Comparison: Placebo vs Spesolimab 'Speso Low' vs Spesolimab 'Speso Medium-low' vs Spesolimab 'Speso Medium-high' vs Spesolimab 'Speso High'; [analysis description as in outcome 1, analysis 5]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.1950, MCP-Mod Logistic model fit — Adjusted for multiplicity; Assumed 20% of maximum effect was achieved at the "low dose", 95% of maximum effect was achieved at "medium high dose"
Statistical Analysis 9: Comparison: Placebo vs Spesolimab 'Speso Low' vs Spesolimab 'Speso Medium-low' vs Spesolimab 'Speso Medium-high' vs Spesolimab 'Speso High'; [analysis description as in outcome 1, analysis 5]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.1681, MCP-Mod Sigmoid Emax model fit — Adjusted for multiplicity; [statistical method as in outcome 1, analysis 9]

4. Secondary Outcome: Palmoplantar Pustulosis Severity Index (PPP SI) Change From Baseline at Week 16
Description: PPP SI change from baseline at Week 16. The PPP SI is based on the severity score of individual components (erythema, pustules, and scaling/desquamation) of PPP ASI assessments. The most severely affected area based on pustules was identified by the investigator at baseline and assessed at all subsequent visits. The PPP SI was calculated by summing up the individual components of PPP ASI assessment (range 0 (best) to 12 (worst)) at each visit for the identified location.
  Least square (LS) means, differences and confidence intervals were estimated by (Restricted maximum likelihood)-based Mixed effect model for repeated measurements (MMRM) including the fixed, categorical effects of treatment at each visit, region and the continuous effect of baseline at each visit as well as random effects of subject. Values post rescue medication or 6 weeks following last study treatment before discontinuation were censored. Unstructured covariance matrix was used.
Time Frame: week 0 (baseline) and week 16.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Placebo | Spesolimab 'Speso Low' | Spesolimab 'Speso Medium-low' | Spesolimab 'Speso Medium-high' | Spesolimab 'Speso High'
Number analyzed (Participants) | 38 | 20 | 21 | 20 | 41
Score on a scale | -2.7 [-3.4 to -2.0] | -3.3 [-4.3 to -2.4] | -3.2 [-4.2 to -2.3] | -3.5 [-4.4 to -2.5] | -2.8 [-3.4 to -2.1]
Statistical Analysis 1: Comparison: Placebo vs Spesolimab 'Speso Low'; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.2812, Mixed Models Analysis; Kenward-Roger was used to estimate denominator degrees of freedom; Difference of adjusted means = -0.7, 95% CI 2-sided [-1.8 to 0.5], Standard Error of Mean 0.6 — Difference was calculated as Speso - placebo
Statistical Analysis 2: Comparison: Placebo vs Spesolimab 'Speso Medium-low'; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.3357, Mixed Models Analysis; Kenward-Roger was used to estimate denominator degrees of freedom; Difference of adjusted means = -0.6, 95% CI 2-sided [-1.7 to 0.6], Standard Error of Mean 0.6 — Difference was calculated as Speso - placebo
Statistical Analysis 3: Comparison: Placebo vs Spesolimab 'Speso Medium-high'; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.1809, Mixed Models Analysis; Kenward-Roger was used to estimate denominator degrees of freedom; Difference of adjusted means = -0.8, 95% CI 2-sided [-2.0 to 0.4], Standard Error of Mean 0.6 — Difference was calculated as Speso - placebo
Statistical Analysis 4: Comparison: Placebo vs Spesolimab 'Speso High'; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.8322, Mixed Models Analysis; Kenward-Roger was used to estimate denominator degrees of freedom; Difference of adjusted means = -0.1, 95% CI 2-sided [-1.1 to 0.9], Standard Error of Mean 0.5 — Difference was calculated as Speso - placebo
Statistical Analysis 5: Comparison: Placebo vs Spesolimab 'Speso Low' vs Spesolimab 'Speso Medium-low' vs Spesolimab 'Speso Medium-high' vs Spesolimab 'Speso High'; [analysis description as in outcome 1, analysis 5]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.4035, MCP-Mod linear model fit — Adjusted for multiplicity
Statistical Analysis 6: Comparison: Placebo vs Spesolimab 'Speso Low' vs Spesolimab 'Speso Medium-low' vs Spesolimab 'Speso Medium-high' vs Spesolimab 'Speso High'; [analysis description as in outcome 1, analysis 5]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.2563, MCP-Mod Emax model fit — Adjusted for multiplicity; Assumed 70% of the maximum effect was achieved at the "low dose" regimen
Statistical Analysis 7: Comparison: Placebo vs Spesolimab 'Speso Low' vs Spesolimab 'Speso Medium-low' vs Spesolimab 'Speso Medium-high' vs Spesolimab 'Speso High'; [analysis description as in outcome 1, analysis 5]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.6810, MCP-Mod Exponential model fit — Adjusted for multiplicity; Assumed 25% of the maximum effect was achieved at the "medium-low dose" regimen
Statistical Analysis 8: Comparison: Placebo vs Spesolimab 'Speso Low' vs Spesolimab 'Speso Medium-low' vs Spesolimab 'Speso Medium-high' vs Spesolimab 'Speso High'; [analysis description as in outcome 1, analysis 5]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.4665, MCP-Mod Logistic model fit — Adjusted for multiplicity; Assumed 20% of maximum effect was achieved at the "low dose", 95% of maximum effect was achieved at "medium high dose"
Statistical Analysis 9: Comparison: Placebo vs Spesolimab 'Speso Low' vs Spesolimab 'Speso Medium-low' vs Spesolimab 'Speso Medium-high' vs Spesolimab 'Speso High'; [analysis description as in outcome 1, analysis 5]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.5565, MCP-Mod Sigmoid Emax model fit — Adjusted for multiplicity; [statistical method as in outcome 1, analysis 9]

5. Secondary Outcome: Number of Patients Achieving a 50% Decrease From Baseline in Palmoplantar Pustulosis Area and Severity Index Score at Week 16 (PPP ASI50)
Description: Number of patients achieving a 50% decrease from baseline in Palmoplantar Pustulosis Area and Severity Index score at week 16 (PPP ASI50). The PPP ASI is an investigator assessment of the extent and severity of palmoplantar pustulosis lesions on the palms and soles in PPP patients. This tool provides a numeric scoring for patients overall PPP disease state, ranging from 0 (best) to 72 (worst). It is a linear combination of the percent of surface area of skin that is affected on the palms and soles of the body and the severity of erythema, pustules, and scaling (desquamation). When (PPP ASI baseline - PPP ASI current)/ PPP ASI baseline * 100% >= 50%, PPP ASI50 = 1.
Time Frame: week 0 (baseline) and week 16
Population: Full Analysis Set (FAS): This patient set includes all patients who were randomised and received at least one dose of study drug and who had a baseline for the primary efficacy endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Spesolimab 'Speso Low' | Spesolimab 'Speso Medium-low' | Spesolimab 'Speso Medium-high' | Spesolimab 'Speso High'
Number analyzed (Participants) | 43 | 22 | 21 | 22 | 44
Participants | 12 | 7 | 10 | 12 | 18
Statistical Analysis 1: Comparison: Placebo vs Spesolimab 'Speso Low'; Test type: Other — Logistic regression with fixed classification effects included treatment and region (Japan vs. Non-Japan). In case 0 event are observed a penalized regression based on the Firth's bias reduction method was used. The estimates from the logistic regression are on the logit scale, the difference in proportions were calculated as the difference between the predicted probabilities in the treatment groups on the original scale; Risk Difference (RD) = 0.042, 95% CI 2-sided [-0.170 to 0.281] — Confidence intervals were calculated using the cumulative distribution function method of Reeve. Difference was calculated as Speso - placebo
Statistical Analysis 2: Comparison: Placebo vs Spesolimab 'Speso Medium-low'; Test type: Other — [test comment as in outcome 5, analysis 1]; Risk Difference (RD) = 0.195, 95% CI 2-sided [-0.048 to 0.432] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Spesolimab 'Speso Medium-high'; Test type: Other — [test comment as in outcome 5, analysis 1]; Risk Difference (RD) = 0.270, 95% CI 2-sided [0.020 to 0.496] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs Spesolimab 'Speso High'; Test type: Other — [test comment as in outcome 5, analysis 1]; Risk Difference (RD) = 0.129, 95% CI 2-sided [-0.067 to 0.314] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs Spesolimab 'Speso Low' vs Spesolimab 'Speso Medium-low' vs Spesolimab 'Speso Medium-high' vs Spesolimab 'Speso High'; [analysis description as in outcome 1, analysis 5]; Test type: Other — Logistic regression estimates were used as input for the MCP-Mod, with fixed classification effects including treatment and region (Japan vs. Non-Japan). In case 0 event are observed a penalized regression based on the Firth's bias reduction method was used. The estimates from the logistic regression are on the logit scale, the difference in proportions were calculated as the difference between the predicted probabilities in the treatment groups on the original scale; p = 0.0613, MCP-Mod linear model fit — Adjusted for multiplicity
Statistical Analysis 6: Comparison: Placebo vs Spesolimab 'Speso Low' vs Spesolimab 'Speso Medium-low' vs Spesolimab 'Speso Medium-high' vs Spesolimab 'Speso High'; [analysis description as in outcome 1, analysis 5]; Test type: Other — [test comment as in outcome 5, analysis 5]; p = 0.0628, MCP-Mod Emax model fit — Adjusted for multiplicity; Assumed 70% of the maximum effect was achieved at the "low dose" regimen
Statistical Analysis 7: Comparison: Placebo vs Spesolimab 'Speso Low' vs Spesolimab 'Speso Medium-low' vs Spesolimab 'Speso Medium-high' vs Spesolimab 'Speso High'; [analysis description as in outcome 1, analysis 5]; Test type: Other — [test comment as in outcome 5, analysis 5]; p = 0.1449, MCP-Mod Exponential model fit — Adjusted for multiplicity; Assumed 25% of the maximum effect was achieved at the "medium-low dose" regimen
Statistical Analysis 8: Comparison: Placebo vs Spesolimab 'Speso Low' vs Spesolimab 'Speso Medium-low' vs Spesolimab 'Speso Medium-high' vs Spesolimab 'Speso High'; [analysis description as in outcome 1, analysis 5]; Test type: Other — [test comment as in outcome 5, analysis 5]; p = 0.0460, MCP-Mod Logistic model fit — Adjusted for multiplicity; Assumed 20% of maximum effect was achieved at the "low dose", 95% of maximum effect was achieved at "medium high dose"
Statistical Analysis 9: Comparison: Placebo vs Spesolimab 'Speso Low' vs Spesolimab 'Speso Medium-low' vs Spesolimab 'Speso Medium-high' vs Spesolimab 'Speso High'; [analysis description as in outcome 1, analysis 5]; Test type: Other — [test comment as in outcome 5, analysis 5]; p = 0.0677, MCP-Mod Sigmoid Emax model fit — Adjusted for multiplicity; [statistical method as in outcome 1, analysis 9]

6. Secondary Outcome: Number of Patients Achieving a 75% Decrease From Baseline in Palmoplantar Pustulosis Area and Severity Index Score at Week 16 (PPP ASI75)
Description: Number of patients achieving a 75% decrease from baseline in Palmoplantar Pustulosis Area and Severity Index score at week 16 (PPP ASI75). The PPP ASI is an investigator assessment of the extent and severity of palmoplantar pustulosis lesions on the palms and soles in PPP patients. This tool provides a numeric scoring for patients overall PPP disease state, ranging from 0 (best) to 72 (worst). It is a linear combination of the percent of surface area of skin that is affected on the palms and soles of the body and the severity of erythema, pustules, and scaling (desquamation). When (PPP ASI baseline - PPP ASI current)/ PPP ASI baseline * 100% >= 75%, PPP ASI75 = 1.
Time Frame: week 0 (baseline) and week 16
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Spesolimab 'Speso Low' | Spesolimab 'Speso Medium-low' | Spesolimab 'Speso Medium-high' | Spesolimab 'Speso High'
Number analyzed (Participants) | 43 | 22 | 21 | 22 | 44
Participants | 3 | 3 | 6 | 4 | 9
Statistical Analysis 1: Comparison: Placebo vs Spesolimab 'Speso Low'; Test type: Other — [test comment as in outcome 5, analysis 1]; Risk Difference (RD) = 0.063, 95% CI 2-sided [-0.069 to 0.256] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Spesolimab 'Speso Medium-low'; Test type: Other — [test comment as in outcome 5, analysis 1]; Risk Difference (RD) = 0.188, 95% CI 2-sided [0.018 to 0.405] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Spesolimab 'Speso Medium-high'; Test type: Other — [test comment as in outcome 5, analysis 1]; Risk Difference (RD) = 0.102, 95% CI 2-sided [-0.042 to 0.303] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs Spesolimab 'Speso High'; Test type: Other — [test comment as in outcome 5, analysis 1]; Risk Difference (RD) = 0.113, 95% CI 2-sided [-0.018 to 0.250] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs Spesolimab 'Speso Low' vs Spesolimab 'Speso Medium-low' vs Spesolimab 'Speso Medium-high' vs Spesolimab 'Speso High'; [analysis description as in outcome 1, analysis 5]; Test type: Other — [test comment as in outcome 5, analysis 5]; p = 0.0536, MCP-Mod linear model fit — Adjusted for multiplicity
Statistical Analysis 6: Comparison: Placebo vs Spesolimab 'Speso Low' vs Spesolimab 'Speso Medium-low' vs Spesolimab 'Speso Medium-high' vs Spesolimab 'Speso High'; [analysis description as in outcome 1, analysis 5]; Test type: Other — [test comment as in outcome 5, analysis 5]; p = 0.0476, MCP-Mod Emax model fit — Adjusted for multiplicity; Assumed 70% of the maximum effect was achieved at the "low dose" regimen
Statistical Analysis 7: Comparison: Placebo vs Spesolimab 'Speso Low' vs Spesolimab 'Speso Medium-low' vs Spesolimab 'Speso Medium-high' vs Spesolimab 'Speso High'; [analysis description as in outcome 1, analysis 5]; Test type: Other — [test comment as in outcome 5, analysis 5]; p = 0.1076, MCP-Mod Exponential model fit — Adjusted for multiplicity; Assumed 25% of the maximum effect was achieved at the "medium-low dose" regimen
Statistical Analysis 8: Comparison: Placebo vs Spesolimab 'Speso Low' vs Spesolimab 'Speso Medium-low' vs Spesolimab 'Speso Medium-high' vs Spesolimab 'Speso High'; [analysis description as in outcome 1, analysis 5]; Test type: Other — [test comment as in outcome 5, analysis 5]; p = 0.0606, MCP-Mod Logistic model fit — Adjusted for multiplicity; Assumed 20% of maximum effect was achieved at the "low dose", 95% of maximum effect was achieved at "medium high dose"
Statistical Analysis 9: Comparison: Placebo vs Spesolimab 'Speso Low' vs Spesolimab 'Speso Medium-low' vs Spesolimab 'Speso Medium-high' vs Spesolimab 'Speso High'; [analysis description as in outcome 1, analysis 5]; Test type: Other — [test comment as in outcome 5, analysis 5]; p = 0.0824, MCP-Mod Sigmoid Emax model fit — Adjusted for multiplicity; [statistical method as in outcome 1, analysis 9]

7. Secondary Outcome: Number of Patients With Palmoplantar Pustulosis Physician Global Assessment (PPP PGA) Clear/Almost Clear (0 or 1) at Week 16
Description: Number of patients with Palmoplantar Pustulosis Physician Global Assessment (PPP PGA) clear/almost clear (0 or 1) at Week 16. The PPP PGA relies on investigator assessment of the patient's skin presentation on the palms and soles. The investigator scored the individual components (erythema, pustules, and scaling/crusting) from 0 (best) to 4 (worst) as clear, almost clear, mild, moderate or severe. PPP PGA categorization is based on the mean of the four individual components.
Time Frame: week 0 (baseline) and week 16
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Spesolimab 'Speso Low' | Spesolimab 'Speso Medium-low' | Spesolimab 'Speso Medium-high' | Spesolimab 'Speso High'
Number analyzed (Participants) | 43 | 22 | 21 | 22 | 44
Participants | 2 | 6 | 4 | 4 | 9
Statistical Analysis 1: Comparison: Placebo vs Spesolimab 'Speso Low'; Test type: Other — [test comment as in outcome 5, analysis 1]; Risk Difference (RD) = 0.211, 95% CI 2-sided [0.040 to 0.422] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Spesolimab 'Speso Medium-low'; Test type: Other — [test comment as in outcome 5, analysis 1]; Risk Difference (RD) = 0.130, 95% CI 2-sided [-0.018 to 0.339] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Spesolimab 'Speso Medium-high'; Test type: Other — [test comment as in outcome 5, analysis 1]; Risk Difference (RD) = 0.125, 95% CI 2-sided [-0.022 to 0.328] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs Spesolimab 'Speso High'; Test type: Other — [test comment as in outcome 5, analysis 1]; Risk Difference (RD) = 0.144, 95% CI 2-sided [0.009 to 0.282] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs Spesolimab 'Speso Low' vs Spesolimab 'Speso Medium-low' vs Spesolimab 'Speso Medium-high' vs Spesolimab 'Speso High'; [analysis description as in outcome 1, analysis 5]; Test type: Other — [test comment as in outcome 5, analysis 5]; p = 0.0333, MCP-Mod linear model fit — Adjusted for multiplicity
Statistical Analysis 6: Comparison: Placebo vs Spesolimab 'Speso Low' vs Spesolimab 'Speso Medium-low' vs Spesolimab 'Speso Medium-high' vs Spesolimab 'Speso High'; [analysis description as in outcome 1, analysis 5]; Test type: Other — [test comment as in outcome 5, analysis 5]; p = 0.0221, MCP-Mod Emax model fit — Adjusted for multiplicity; Assumed 70% of the maximum effect was achieved at the "low dose" regime
Statistical Analysis 7: Comparison: Placebo vs Spesolimab 'Speso Low' vs Spesolimab 'Speso Medium-low' vs Spesolimab 'Speso Medium-high' vs Spesolimab 'Speso High'; [analysis description as in outcome 1, analysis 5]; Test type: Other — [test comment as in outcome 5, analysis 5]; p = 0.0707, MCP-Mod Exponential model fit — Adjusted for multiplicity; Assumed 25% of the maximum effect was achieved at the "medium-low dose" regimen
Statistical Analysis 8: Comparison: Placebo vs Spesolimab 'Speso Low' vs Spesolimab 'Speso Medium-low' vs Spesolimab 'Speso Medium-high' vs Spesolimab 'Speso High'; [analysis description as in outcome 1, analysis 5]; Test type: Other — [test comment as in outcome 5, analysis 5]; p = 0.0578, MCP-Mod Logistic model fit — Adjusted for multiplicity; Assumed 20% of maximum effect was achieved at the "low dose", 95% of maximum effect was achieved at "medium high dose"
Statistical Analysis 9: Comparison: Placebo vs Spesolimab 'Speso Low' vs Spesolimab 'Speso Medium-low' vs Spesolimab 'Speso Medium-high' vs Spesolimab 'Speso High'; [analysis description as in outcome 1, analysis 5]; Test type: Other — [test comment as in outcome 5, analysis 5]; p = 0.0771, MCP-Mod Sigmoid Emax model fit — Adjusted for multiplicity; [statistical method as in outcome 1, analysis 9]

8. Secondary Outcome: Number of Patients With Palmoplantar Pustulosis Physician Global Assessment (PPP PGA) Pustules Clear/Almost Clear (0 or 1) at Week 16
Description: Number of patients with Palmoplantar Pustulosis Physician Global Assessment (PPP PGA) pustules clear/almost clear (0 or 1) at Week 16. The PPP PGA relies on investigator assessment of the patient's skin presentation on the palms and soles. The investigator scored the pustules from 0 (best) to 4 (worst) as clear, almost clear, mild, moderate or severe.
Time Frame: week 0 (baseline) and week 16
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Spesolimab 'Speso Low' | Spesolimab 'Speso Medium-low' | Spesolimab 'Speso Medium-high' | Spesolimab 'Speso High'
Number analyzed (Participants) | 43 | 22 | 21 | 22 | 44
Participants | 5 | 7 | 6 | 8 | 14
Statistical Analysis 1: Comparison: Placebo vs Spesolimab 'Speso Low'; Test type: Other — [test comment as in outcome 5, analysis 1]; Risk Difference (RD) = 0.202, 95% CI 2-sided [-0.005 to 0.427] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Spesolimab 'Speso Medium-low'; Test type: Other — [test comment as in outcome 5, analysis 1]; Risk Difference (RD) = 0.170, 95% CI 2-sided [-0.032 to 0.401] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Spesolimab 'Speso Medium-high'; Test type: Other — [test comment as in outcome 5, analysis 1]; Risk Difference (RD) = 0.248, 95% CI 2-sided [0.032 to 0.471] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs Spesolimab 'Speso High'; Test type: Other — [test comment as in outcome 5, analysis 1]; Risk Difference (RD) = 0.202, 95% CI 2-sided [0.024 to 0.367] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs Spesolimab 'Speso Low' vs Spesolimab 'Speso Medium-low' vs Spesolimab 'Speso Medium-high' vs Spesolimab 'Speso High'; [analysis description as in outcome 1, analysis 5]; Test type: Other — [test comment as in outcome 5, analysis 5]; p = 0.0158, MCP-Mod linear model fit — Adjusted for multiplicity
Statistical Analysis 6: Comparison: Placebo vs Spesolimab 'Speso Low' vs Spesolimab 'Speso Medium-low' vs Spesolimab 'Speso Medium-high' vs Spesolimab 'Speso High'; [analysis description as in outcome 1, analysis 5]; Test type: Other — [test comment as in outcome 5, analysis 5]; p = 0.0120, MCP-Mod Emax model fit — Adjusted for multiplicity; Assumed 70% of the maximum effect was achieved at the "low dose" regimen
Statistical Analysis 7: Comparison: Placebo vs Spesolimab 'Speso Low' vs Spesolimab 'Speso Medium-low' vs Spesolimab 'Speso Medium-high' vs Spesolimab 'Speso High'; [analysis description as in outcome 1, analysis 5]; Test type: Other — [test comment as in outcome 5, analysis 5]; p = 0.0429, MCP-Mod Exponential model fit — Adjusted for multiplicity; Assumed 25% of the maximum effect was achieved at the "medium-low dose" regimen
Statistical Analysis 8: Comparison: Placebo vs Spesolimab 'Speso Low' vs Spesolimab 'Speso Medium-low' vs Spesolimab 'Speso Medium-high' vs Spesolimab 'Speso High'; [analysis description as in outcome 1, analysis 5]; Test type: Other — [test comment as in outcome 5, analysis 5]; p = 0.0229, MCP-Mod Logistic model fit — Adjusted for multiplicity; Assumed 20% of maximum effect was achieved at the "low dose", 95% of maximum effect was achieved at "medium high dose"
Statistical Analysis 9: Comparison: Placebo vs Spesolimab 'Speso Low' vs Spesolimab 'Speso Medium-low' vs Spesolimab 'Speso Medium-high' vs Spesolimab 'Speso High'; [analysis description as in outcome 1, analysis 5]; Test type: Other — [test comment as in outcome 5, analysis 5]; p = 0.0300, MCP-Mod Sigmoid Emax model fit — Adjusted for multiplicity; [statistical method as in outcome 1, analysis 9]

9. Secondary Outcome: The Percentage Change in Palmoplantar Pustulosis Area and Severity Index (PPP ASI) at Week 52 From Baseline
Description: The percentage change in PPP ASI at Week 52 from baseline. The PPP ASI is an investigator assessment of the extent and severity of palmoplantar pustulosis lesions on the palms and soles in PPP patients. This tool provides a numeric scoring for patients overall PPP disease state, ranging from 0 (best) to 72 (worst). It is a linear combination of the percent of surface area of skin that is affected on the palms and soles of the body and the severity of erythema, pustules, and scaling (desquamation).
  LS means, differences and confidence intervals were estimated by (Restricted maximum likelihood)-based MMRM including the fixed, categorical effects of treatment at each visit, region and the continuous effect of baseline at each visit as well as random effects of subject. Values post rescue medication or 6 weeks following last study treatment before discontinuation were censored. Unstructured covariance matrix was used.
Time Frame: week 0 (baseline) and week 52
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of change in PPP ASI
Arm/Group | Placebo & Spesolimab | Spesolimab 'Speso Low' | Spesolimab 'Speso Medium-low' | Spesolimab 'Speso Medium-high' | Spesolimab 'Speso High'
Number analyzed (Participants) | 32 | 19 | 18 | 17 | 32
Percentage of change in PPP ASI | -54.6 [-65.8 to -43.3] | -73.3 [-87.9 to -58.6] | -73.8 [-89.1 to -58.6] | -81.2 [-96.4 to -66.1] | -60.0 [-70.9 to -49.2]
Statistical Analysis 1: Comparison: Placebo & Spesolimab vs Spesolimab 'Speso Low'; Test type: Other — MMRM included 'baseline' as a continuous covariate, and 'visit', 'treatment', 'region' (stratification according to Japan vs. non-Japan), 'visit*treatment' and 'visit*baseline' interaction as fixed effects as well as the random 'subject' effect. Covariance structure= Unstructured; Difference of adjusted means = -18.7, 95% CI 2-sided [-37.2 to -0.2], Standard Error of Mean 9.3 — Difference was calculated as Speso - placebo
Statistical Analysis 2: Comparison: Placebo & Spesolimab vs Spesolimab 'Speso Medium-low'; Test type: Other — [test comment as in outcome 9, analysis 1]; Difference of adjusted means = -19.3, 95% CI 2-sided [-38.3 to -0.2], Standard Error of Mean 9.6 — Difference was calculated as Speso - placebo
Statistical Analysis 3: Comparison: Placebo & Spesolimab vs Spesolimab 'Speso Medium-high'; Test type: Other — [test comment as in outcome 9, analysis 1]; Difference of adjusted means = -26.6, 95% CI 2-sided [-45.5 to -7.8], Standard Error of Mean 9.5 — Difference was calculated as Speso - placebo
Statistical Analysis 4: Comparison: Placebo & Spesolimab vs Spesolimab 'Speso High'; Test type: Other — [test comment as in outcome 9, analysis 1]; Difference of adjusted means = -5.4, 95% CI 2-sided [-21.1 to 10.2], Standard Error of Mean 7.9 — Difference was calculated as Speso - placebo

ADVERSE EVENTS:
Time Frame: Adverse events: first until the last day of study drug administration + 112 days, up to 68 weeks.
Description: Safety analysis set (SAF): This patient set includes all patients who were randomised and received at least one dose of study drug.
Groups:
- Spesolimab Post Placebo: Subcutaneous injections of Spesolimab starting at week 16, for a total treatment time until week 52.
Arm/Group | Placebo | Spesolimab Post Placebo | Spesolimab 'Speso Low' | Spesolimab 'Speso Medium-low' | Spesolimab 'Speso Medium-high' | Spesolimab 'Speso High'
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/38 | 0/22 | 0/21 | 0/22 | 0/44
Serious Adverse Events (participants affected / at risk) | 2/43 | 3/38 | 3/22 | 5/21 | 3/22 | 3/44
Other Adverse Events (participants affected / at risk) | 24/43 | 22/38 | 17/22 | 17/21 | 17/22 | 31/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=43) | Spesolimab Post Placebo (N=38) | Spesolimab 'Speso Low' (N=22) | Spesolimab 'Speso Medium-low' (N=21) | Spesolimab 'Speso Medium-high' (N=22) | Spesolimab 'Speso High' (N=44)
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0
Retinal artery embolism (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Palmoplantar pustulosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=43) | Spesolimab Post Placebo (N=38) | Spesolimab 'Speso Low' (N=22) | Spesolimab 'Speso Medium-low' (N=21) | Spesolimab 'Speso Medium-high' (N=22) | Spesolimab 'Speso High' (N=44)
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 3 | 2 | 2 | 1
Injection site erythema (General disorders) | 0 | 2 | 3 | 1 | 4 | 3
Injection site pain (General disorders) | 3 | 2 | 0 | 3 | 1 | 1
Injection site reaction (General disorders) | 0 | 4 | 3 | 5 | 5 | 20
Pyrexia (General disorders) | 0 | 0 | 1 | 2 | 0 | 0
Nasopharyngitis (Infections and infestations) | 5 | 3 | 3 | 2 | 2 | 4
Rhinitis (Infections and infestations) | 3 | 0 | 1 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 2 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 3 | 0 | 1 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 3
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 4
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 4 | 3 | 0 | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 1 | 2 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0 | 0 | 0
Pustulotic arthro-osteitis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 2 | 2
Headache (Nervous system disorders) | 1 | 3 | 2 | 0 | 2 | 5
Insomnia (Psychiatric disorders) | 3 | 0 | 1 | 0 | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 3 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 2 | 2 | 6 | 2 | 1 | 0
Palmoplantar pustulosis (Skin and subcutaneous tissue disorders) | 4 | 0 | 1 | 1 | 1 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 0 | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-04-03): https://cdn.clinicaltrials.gov/large-docs/18/NCT04015518/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-22): https://cdn.clinicaltrials.gov/large-docs/18/NCT04015518/SAP_001.pdf